CLINICAL TRIAL: NCT00253786
Title: Study for the Effectiveness of Intensive Therapy for Diabetic Nephropathy in Unblinded, Randomized Intergroup Comparison Study.
Brief Title: Study for the Effectiveness of Intensive Therapy Aiming at a Remission of Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okayama University (Other)
Responsible Party: Principal Investigator, Kenichi Shikata, Professor, Okayama University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNETT-Japan
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Nephropathy
Keywords: diabetes; nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases | interventions — Standard of Care

ARMS (4):
- Intensive multifactorial therapy (Protocol A) (Experimental): Protocol A: serum creatinine <1.2 mg/dl in male and <1.0 mg/dl in female.
  Interventions: Other: Intensive multifactorial therapy
- Standard therapy (Protocol A) (Active Comparator): Protocol A: serum creatinine <1.2 mg/dl in male and <1.0 mg/dl in female.
  Interventions: Other: Standard therapy
- Intensive multifactorial therapy (Protocol B) (Experimental): Protocol B: serum creatinine: 1.2-2.5 mg/dl in male and 1.0-2.5 mg/dl in female.
  Interventions: Other: Intensive multifactorial therapy
- Standard therapy (Protocol B) (Active Comparator): Protocol B: serum creatinine: 1.2-2.5 mg/dl in male and 1.0-2.5 mg/dl in female.
  Interventions: Other: Standard therapy

INTERVENTIONS:
Other: Intensive multifactorial therapy — Blood glucose control: HbA1c < 6.2% Blood pressure control: SBP < 125 mmHg, DBP: < 75 mmHg Lipid profile: T-cho < 180 mg/dl, LDL-cho < 100 mg/dl, HDL-cho >40 mg/dl Dietary intervention: TDEI < 30 kcal/kg/day, sodium < 5 g/day, protein < 0.8 g/kg/day Pharmacological intervention: ACE-Is or ARBs, HMG-CoA reductase inhibitors, multivitamins Instruction by co-medicals: Taking medicines, smoking cessation, nutrition care
  Arms: Intensive multifactorial therapy (Protocol A); Intensive multifactorial therapy (Protocol B)
Other: Standard therapy — Blood glucose control: HbA1c < 6.9% Blood pressure control: SBP < 130 mmHg, DBP: < 80 mmHg Lipid profile: T-cho < 200 mg/dl, LDL-cho < 120 mg/dl, HDL-cho >40 mg/dl, Dietary intervention: TDEI < 25-30 kcal/kg/day, sodium < 6 g/day, protein < 1.0 g/kg/day Pharmacological intervention: No restrictions (continuing prior therapy) Instruction by co-medicals: No restrictions (continuing prior therapy)
  Arms: Standard therapy (Protocol A); Standard therapy (Protocol B)

SUMMARY:
Study for the effectiveness of intensive therapy aiming at the remission of diabetic nephropathy

DETAILED DESCRIPTION:
Study for the effectiveness of intensive therapy for diabetic nephropathy in unblinded, randomized intergroup comparison study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes
2. Urinary albumin-to-creatinine ratio: >=300 mg/g creatinine twice in the first morning urine sample
3. Serum creatinine level: =<2.5 mg/dl
4. Patients aged 20-75 years

Exclusion Criteria:

1. Type 1 diabetes
2. Hereditary diabetes or secondary diabetes
3. Non-diabetic nephropathy
4. Familial hypercholesterolemia
5. Secondary hypertension
6. Unstable angina pectoris or history of myocardial infarction/stroke within 6 months prior to consent acquisition
7. Malignant tumor or life threatening disease
8. History of angioedema
9. Patients undergoing LDL apheresis
10. Biliary system obstruction or severe liver injury
11. Liver dysfunction
12. Allergy for ACE-Is, ARBs or HMG-CoA reductase inhibitors
13. Pregnant or nursing patients
14. Others: patients who are not suitable for this trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2005-11-11 (Actual); Primary Completion 2014-11-27 (Actual); Study Completion 2014-11-27 (Actual)

PRIMARY OUTCOMES:
Urinary protein/creatinine ratio (in the first morning urine sample) in Protocol A | 5 years
Composite endpoint of time to first occurrence of (1) Doubling of serum creatinine, (2) Need for chronic dialysis or renal transplantation, or (3) Death in Protocol B | 5 years

SECONDARY OUTCOMES:
GFR in Protocol A | 5 years
Cardiovascular event in Protocol A | 5 years
Progression of retinopathy in Protocol A | 5 years
Urinary albumin/creatinine ratio in Protocol A | 5 years
Proteinuria (24 h collection sample) in Protocol A | 5 years
GFR in Protocol B | 5 years
Cardiovascular event in Protocol B | 5 years
Progression of retinopathy in Protocol B | 5 years
Urinary albumin/creatinine ratio in Protocol B | 5 years
Urinary protein/creatinine ratio in Protocol B | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Makino, M.D., Principal Investigator — Okayama University, Graduate School of Medicine, Dentistry and Pharmaceutical Sciences
Locations (1):
- Okayama University Hospital, Okayama, Japan

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Hodson EM, Cooper TE. Altered dietary salt intake for preventing diabetic kidney disease and its progression. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD006763. doi: 10.1002/14651858.CD006763.pub3. PMID 36645291